CLINICAL TRIAL: NCT00383149
Title: A Phase II, Open Label Trial of Ixabepilone Plus Cetuximab as First Line Therapy for Metastatic Pancreatic Cancer
Brief Title: A Phase II, Trial of Ixabepilone Plus Cetuximab as First Line Therapy for Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-116
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ixabepilone; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone plus Cetuximab (Experimental): All participants were administered ixabepilone at a starting dose of 32 mg/m^2 as a 3-hour intravenous (IV) infusion every 3 weeks. In addition, all participants were administered an initial dose of cetuximab (400 mg/m^2 IV over 2 hours) followed by a weekly lower dose (250 mg/m^2 IV over 1 hour).
  Interventions: Drug: Ixabepilone; Drug: Cetuximab

INTERVENTIONS:
Drug: Ixabepilone — Intravenous Infusion (IV), 32 mg/m^2 every 21 days.
  Other Names: IXEMPRA®; Erbitux®; BMS-247550; BMS-564717
Drug: Cetuximab — Initial dose of 400 mg/m^2 intravenous (IV) over 2 hours) followed by a weekly lower dose of 250 mg/m^2 IV over 1 hour.

SUMMARY:
The purpose of this clinical research study is to learn if ixabepilone plus cetuximab improves survival when given as 1st line chemotherapy in subjects with metastatic pancreatic cancer compared to historical data. The safety of this combination treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of pancreatic adenocarcinoma (locally advanced disease that is not surgically resectable, or distant metastatic disease)
* Participants must have measurable disease as per Response Evaluation Criteria In Solid Tumors (RECIST) guidelines
* Participants must not have received prior chemotherapy, immunotherapy or chemoradiotherapy for advanced pancreas cancer
* Karnofsky performance status (KPS) of 70-100
* Adequate hematologic, hepatic and renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Georgetn Univ Lombardi Can Ctr, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - University Of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 58 participants enrolled, 4 were never treated.
Groups:
- Ixabepilone + Cetuximab: All participants were administered ixabepilone at a starting dose of 32 mg/m^2 as a 3-hour intravenous (IV) infusion every 3 weeks. In addition, all participants were administered an initial dose of cetuximab (400 mg/m^2 IV over 2 hours) followed by a weekly lower dose (250 mg/m^2 IV over 1 hour).
Period: Overall Study
Arm/Group | Ixabepilone + Cetuximab
Started | 54
Completed | 0
Not Completed | 54
Not completed — Adverse Event not Related to Study Drug | 3
Not completed — Death | 2
Not completed — Disease Progression | 38
Not completed — Lost to Follow-up | 1
Not completed — Other | 1
Not completed — Study Drug Toxicity | 4
Not completed — Request to Discontinue Treatment | 4
Not completed — Participant Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 63.0 [47.0 to 84.0]
Age, Customized [Number; unit: participants]
  Age Greater than, equal to 65 years | 22
  Age less than 65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Surviving at 6 Months
Description: The percentage of participants surviving at 6 months was defined as the number of treated participants who had not died prior to 6 months from the date of their first dose divided by the total number of treated participants.
Time Frame: From time of first dose of study drug through 6 months
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab. Participants who did not die prior to 6 months but dropped out of the study were not included in the numerator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
percentage of participants | 57.4 [43.2 to 70.8]

2. Secondary Outcome: Best Overall Tumor Response
Description: Tumor response was assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)= disappearance of all non-target lesions, Partial Response (PR)= at least 30% reduction in the sum of the longest diameter (LD) of all target lesions in reference to the baseline sum LD; Stable Disease (SD)= neither PR nor progressive disease (PD) criteria were met; PD = at least 20% increase in the sum of the LD of all target lesions, taking as reference the smallest sum LD recorded at or following baseline.
Time Frame: From time of first dose of study until 16.49 months (longest period for participant between first dose and documented disease progression)
Population: Response-evaluable participants; all participants with measurable disease who received at least one dose of ixabepilone or cetuximab and who had at least one on-treatment tumor assessment.
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 31
participants
  Participants with Complete Response | 0
  Participants with Partial Response | 4
  Participants with Stable Disease | 24
  Participants with Progressive Disease | 2
  Participants with Response Unable to be Determined | 1

3. Secondary Outcome: Percentage of Participants With Objective Tumor Response
Description: Percentage of participants with objective tumor response was determined by the number of participants with PR or CR divided by the total number of response-evaluable participants. Tumor response was assessed according RECIST criteria: PR=at least 30% reduction in the sum of the LD of all target lesions in reference to the baseline sum LD, CR=Disappearance of all non-target lesions.
Time Frame: From time of first dose of study until 16.49 months (longest period for participant between first dose and documented disease progression
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 31
percentage of participants | 12.9 [3.6 to 29.8]

4. Secondary Outcome: Median Progression Free Survival Time
Description: Progression-Free Survival (PFS) time was defined as the time, in months, from the first dosing date until the date of disease progression or death from any cause.
Time Frame: as for outcome 3
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab. Participants without disease progression or death were censored at the last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
months | 3.9 [2.6 to 4.4]

5. Secondary Outcome: Median Overall Survival Time
Description: Overall survival time was defined as the time in months from the first dosing date to the date of death.
Time Frame: From the first dosing date until death (last reported death was 21 months after first dose).
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab. Participants without a reported date of death were censored at the last known alive date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
months | 7.6 [5.5 to 12.2]

6. Secondary Outcome: Median Duration of Response
Description: Duration of response was defined as the number of months from when measurement criteria were first met for CR or PR (whichever was recorded first) until the first date of disease progression or death. Complete Response (CR)= disappearance of all non-target lesions, Partial Response (PR)= at least 30% reduction in the sum of the longest diameter (LD) of all target lesions in reference to the baseline sum LD.
Time Frame: From first date recorded for CR or PR until the first date of disease progression or death (last participant with tumor response progressed 6.5 months after documented response).
Population: Response-evaluable participants whose best response was PR or CR. Participants without disease progression or death were censored at the last tumor assessment date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 4
months | 5.7 [2.8 to 6.3]

7. Secondary Outcome: Median Time to Response
Description: Time to response was defined as the number of weeks from first dose of study therapy (ixabepilone or cetuximab) until measurement criteria were first met for PR or CR, whichever status was recorded first. Complete Response (CR)= disappearance of all non-target lesions, Partial Response (PR)= at least 30% reduction in the sum of the longest diameter (LD) of all target lesions in reference to the baseline sum LD.
Time Frame: Time from first dose of study therapy until first date of PR or CR. Maximum time to response was 19 months.
Population: Response-evaluable participants whose best response was PR or CR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 4
weeks | 8.8 [5.1 to 19.0]

8. Secondary Outcome: Number of Participants With Death Within 30 Days of Last Dose, Any Serious Adverse Event (SAE), Any Adverse Event (AE) Leading to Discontinuation (DC), or Any Treatment-related AEs By Common Terminology Criteria Version 3.0 (CTC v3) Grade (Gr)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition not necessarily having a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization/causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, or is an important medical event.
Time Frame: From the time of first dose of study drug to ≤30 days after the end of the last dose of study drug or until resolution of study drug-related toxicity.
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab. The 53 participants reporting treatment-related AEs included 1 additional participant who also developed Grade 5 viscous intestinal perforation, which was also captured under death within 30 days of last dose category.
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
participants
  All deaths within 30 days of last dose | 7
  Any SAE | 32
  Gr 2 (moderate) AE leading to DC | 2
  Gr 3 (severe) AE leading to DC | 9
  Gr 4 (life-threatening) AE leading to DC | 3
  All AEs leading to DC | 14
  Gr 1 (mild) treatment-related AE | 4
  Gr 2 (moderate) treatment-related AE | 13
  Gr 3 (severe) treatment-related AE | 25
  Gr 4 (life-threatening) treatment-related AE | 10
  Gr 5 (death) treatment-related AE | 1
  All treatment-related AEs | 53

9. Secondary Outcome: Number of Participants With Most Common Treatment-related Nonhematologic AE (>25%) By CTC v3 Grade (Gr)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition not necessarily having a causal relationship with this treatment. Acneform rash and peripheral neuropathy were captured by multiple MedDRA preferred terms. Acneform rash included rash, rash pustular, and rash pruritic preferred terms. Peripheral neuropathy included neuromuscular toxicity, peripheral motor neuropathy, and peripheral sensorimotor neuropathy preferred terms.
Time Frame: as for outcome 8
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab.
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
participants
  Gr 1 (mild) acneform rash | 21
  Gr 2 (moderate) acneform rash | 13
  Gr 3 (severe) acneform rash | 1
  All acneform rash | 35
  Gr 1 (mild) fatigue | 8
  Gr 2 (moderate) fatigue | 13
  Gr 3 (severe) fatigue | 8
  Gr 4 (life-threatening) fatigue | 1
  All fatigue | 30
  Gr 1 (mild) alopecia | 13
  Gr 2 (moderate) alopecia | 12
  All alopecia | 25
  Gr 1 (mild) nausea | 13
  Gr 2 (moderate) nausea | 6
  Gr 3 (severe) nausea | 3
  All nausea | 22
  Gr 1 (mild) diarrhea | 11
  Gr 2 (moderate) diarrhea | 4
  Gr 3 (severe) diarrhea | 1
  Gr 4 (life-threatening) diarrhea | 2
  All diarrhea | 18
  Gr 1 (mild) vomiting | 12
  Gr 2 (moderate) vomiting | 2
  Gr 3 (severe) vomiting | 3
  All vomiting | 17
  Gr 1 (mild) peripheral neuropathy | 12
  Gr 2 (moderate) peripheral neuropathy | 1
  Gr 3 (severe) peripheral neuropathy | 3
  All peripheral neuropathy | 16
  Gr 1 (mild) hypomagnesemia | 7
  Gr 2 (moderate) hypomagnesemia | 4
  Gr 3 (severe) hypomagnesemia | 1
  Gr 4 (life-threatening) hypomagnesemia | 3
  All hypomagnesemia | 15

10. Secondary Outcome: Number of Participants With Hematology, Liver Function, and Renal Laboratory Abnormalities By CTC v3 Grade (Gr)
Description: Laboratory results were graded according to CTC v 3.0. Hematology laboratory evaluations included absolute neutrophil count (ANC), white blood cell count (WBC), platelets (PLT), and hemoglobin (HGB). Liver function laboratory evaluations included alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin. Renal function laboratory evaluation included creatinine.
Time Frame: as for outcome 8
Population: Treated participants; all participants who received at least one dose of ixabepilone or cetuximab. n= number of participants with laboratory data available
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 54
participants
  Gr 0 (no abnormality) WBC, n=51 | 12
  Gr 1 (mild) WBC, n=51 | 9
  Gr 2 (moderate) WBC, n=51 | 9
  Gr 3 (severe) WBC, n=51 | 17
  Gr 4 (life-threatening) WBC, n=51 | 4
  Gr 1-4 WBC, n=51 | 39
  Gr 3-4 WBC, n=51 | 21
  Gr 0 (no abnormality) ANC, n=50 | 12
  Gr 1 (mild) ANC, n=50 | 8
  Gr 2 (moderate) ANC, n=50 | 12
  Gr 3 (severe) ANC, n=50 | 10
  Gr 4 (life-threatening) ANC, n=50 | 8
  Gr 1-4 ANC, n=50 | 38
  Gr 3-4 ANC, n=51 | 18
  Gr 0 (no abnormality) platelet count, n=51 | 29
  Gr 1 (mild) platelet count, n=51 | 18
  Gr 2 (moderate) platelet count, n=51 | 4
  Gr 1-4 platelet count, n=51 | 2
  Gr 0 (no abnormality) HGB, n=51 | 3
  Gr 1 (mild) HGB, n=51 | 28
  Gr 2 (moderate) HGB, n=51 | 18
  Gr 3 (severe) HGB, n=51 | 2
  Gr 1-4 HGB, n=51 | 48
  Gr 3-4 HGB, n=51 | 2
  Gr 0 (no abnormality) ALT, n=46 | 31
  Gr 1 (mild) ALT, n=46 | 10
  Gr 2 (moderate) ALT, n=46 | 3
  Gr 3 (severe) ALT, n=46 | 2
  Gr 1-4 ALT, n=46 | 15
  Gr 3-4 ALT, n=46 | 2
  Gr 0 (no abnormality) AST, n=47 | 28
  Gr 1 (mild) AST, n=47 | 17
  Gr 3 (severe) AST, n=47 | 2
  Gr 1-4 AST, n=47 | 19
  Gr 3-4 AST, n=47 | 2
  Gr 0 (no abnormality) alkaline phosphatase, n=47 | 18
  Gr 1 (mild) alkaline phosphatase, n=47 | 20
  Gr 2 (moderate) alkaline phosphatase, n=47 | 5
  Gr 3 (severe) alkaline phosphatase, n=47 | 4
  Gr 1-4 alkaline phosphatase, n=47 | 29
  Gr 3-4 alkaline phosphatase, n=47 | 4
  Gr 0 (no abnormality) total bilirubin, n=48 | 42
  Gr 1 (mild) total bilirubin, n=48 | 1
  Gr 2 (moderate) total bilirubin, n=48 | 1
  Gr 3 (severe) total bilirubin, n=48 | 4
  Gr 1-4 total bilirubin, n=48 | 6
  Gr 3-4 total bilirubin, n=48 | 4
  Gr 0 (no abnormality) creatinine, n=48 | 45
  Gr 1 (mild) creatinine, n=48 | 3
  Gr 1-4 creatinine, n=48 | 3

11. Secondary Outcome: Number of Participants With Dose Reduction, Dose Delay, or Dose Interruption
Description: Dose reduction of ixabepilone and/or cetuximab due to toxicity was permitted for participants deriving benefit from therapy. Each drug could be dose modified independently of the others. Participants unable to start a cycle due to unacceptable toxicity related to ixabepilone or cetuximab could have therapy delayed for up to 4 weeks. If toxicities prevented the administration of ixabepilone or cetuximab therapy, participants continued receiving the other therapy as scheduled. A dose interruption for ixabepilone or cetuximab was defined as any interruption during the infusion period.
Time Frame: From the first dosing date of Cycle 1 until the last dosing date of the last cycle. Last dosing cycle for a participant was Cycle 21.
Population: Since the combination of ixabepilone and cetuximab tested in this trial failed to meet the primary objective of sufficiently improving 6-month survival rate relative to historical control in participants with metastatic pancreatic cancer, dose modification data were collected but not summarized.
Groups:
- Ixabepilone: All participants were administered ixabepilone at a starting dose of 32 mg/m^2 as a 3-hour intravenous (IV) infusion every 3 weeks.
- Cetuximab: All participants were administered an initial dose of cetuximab (400 mg/m^2 IV over 2 hours) followed by a weekly lower dose (250 mg/m^2 IV over 1 hour).
Arm/Group | Ixabepilone | Cetuximab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Baseline Epidermal Growth Factor Receptor (EGFR) Tumor Expression
Description: EGFR expression was evaluated by means of an immunohistochemical assay using tumor tissue collected prior to receiving first dose.
Time Frame: Baseline
Population: Tissue was available for a small proportion of patients and only 1 out of 11 was EGFR positive, hence EFGR expression analysis was not performed.
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in FHSI-8 Total Score by Time-point
Description: The FHSI-8 includes eight items representing pancreatic-related symptoms; each symptom is rated by participants on a scale of from 0 to 4. The FHSI-8 total score ranges in value from 0 to 32, with higher scores representing fewer symptoms and lower scores representing more symptoms. Scoring of the FHSI-8 was to be conducted according to the Functional Assessment of Chronic Illness Therapy (FACIT) manual. The symptom assessment was to include treated participants who had baseline measurement and at least one on-study measurement of FHSI-8 questionnaire.
Time Frame: Baseline, Week 3, Week 6, Week 9, Week 12, Week 12, Week 18, Week 24 and every 3 weeks through end of study (participant death/withdrawal from study)
Population: Since the combination of ixabepilone and cetuximab tested in this trial failed to meet the primary objective of sufficiently improving 6-month survival rate relative to historical control in participants with metastatic pancreatic cancer, FHSI-8 score data were collected but not summarized.
Arm/Group | Ixabepilone + Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ixabepilone + Cetuximab
Serious Adverse Events (participants affected / at risk) | 32/54
Other Adverse Events (participants affected / at risk) | 49/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone + Cetuximab (N=54)
WEIGHT DECREASED (Investigations) | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
HYPOTENSION (Vascular disorders) | 6
DEEP VEIN THROMBOSIS (Vascular disorders) | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
CHOLANGITIS (Hepatobiliary disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 3
ANAPHYLACTIC REACTION (Immune system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
NAUSEA (Gastrointestinal disorders) | 3
ASCITES (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 2
STOMATITIS (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
ABDOMINAL MASS (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
BACTERAEMIA (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
LIVER ABSCESS (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 5
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
CHILLS (General disorders) | 1
PYREXIA (General disorders) | 3
VISCERAL OEDEMA (General disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone + Cetuximab (N=54)
WEIGHT DECREASED (Investigations) | 11
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6
HYPOTENSION (Vascular disorders) | 8
ANXIETY (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 9
DEPRESSION (Psychiatric disorders) | 6
HYPERSENSITIVITY (Immune system disorders) | 5
HEADACHE (Nervous system disorders) | 5
DIZZINESS (Nervous system disorders) | 9
DYSGEUSIA (Nervous system disorders) | 3
PARAESTHESIA (Nervous system disorders) | 5
NEUROPATHY PERIPHERAL (Nervous system disorders) | 4
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6
NAUSEA (Gastrointestinal disorders) | 25
ASCITES (Gastrointestinal disorders) | 6
VOMITING (Gastrointestinal disorders) | 18
DIARRHOEA (Gastrointestinal disorders) | 22
FLATULENCE (Gastrointestinal disorders) | 8
STOMATITIS (Gastrointestinal disorders) | 8
CONSTIPATION (Gastrointestinal disorders) | 20
ABDOMINAL PAIN (Gastrointestinal disorders) | 17
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4
PARONYCHIA (Infections and infestations) | 4
URINARY TRACT INFECTION (Infections and infestations) | 4
DYSURIA (Renal and urinary disorders) | 4
ANOREXIA (Metabolism and nutrition disorders) | 17
DEHYDRATION (Metabolism and nutrition disorders) | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 17
ANAEMIA (Blood and lymphatic system disorders) | 14
LEUKOPENIA (Blood and lymphatic system disorders) | 8
LYMPHOPENIA (Blood and lymphatic system disorders) | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 11
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 25
DRY SKIN (Skin and subcutaneous tissue disorders) | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 4
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 29
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
CHILLS (General disorders) | 3
FATIGUE (General disorders) | 34
PYREXIA (General disorders) | 9
ASTHENIA (General disorders) | 5
OEDEMA PERIPHERAL (General disorders) | 7
MUCOSAL INFLAMMATION (General disorders) | 9

LIMITATIONS AND CAVEATS:
Study CA163-116 was completed; however, the combination tested in this trial failed to meet the primary objective to demonstrate a 6-month survival rate greater than 50% in participants with metastatic pancreatic cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.